CLINICAL TRIAL: NCT04398667
Title: A European Non-interventional Study to Understand the Criteria Used and the Time Required for the Clinical Diagnosis in Participants With Refractory Epilepsies Associated With Developmental Delay
Brief Title: European Non-interventional Study on Refractory Epilepsy With Developmental Delay
Status: Terminated | Type: Observational
Why Stopped: The clinical research organization went out of business.
Sponsor: Zogenix, Inc. (Industry)
Collaborators: Zogenix International Limited, Inc., a subsidiary of Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: 915-ENSURED
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Refractory Epilepsy; Development Delay
Keywords: Observational; Retrospective
MeSH Terms: conditions — Drug Resistant Epilepsy; Learning Disabilities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multinational, multicentre, non-interventional, retrospective data collection (manual Medical Chart Review).

DETAILED DESCRIPTION:
This is a multinational, multicentre, non-interventional, retrospective data collection (manual Medical Chart Review). The identified local site staff (or trained independent data abstractors, if requested by the site) will review the medical records of all participants meeting the eligibility criteria, who have provided a signed inform consent form (ICF) for data collection and analysis. For participants who are less than 18 years of age, in addition to the assent form being signed by the participant, an informed consent would be obtained from parental or legally authorized representative.

In line with the retrospective nature of the study: there is no assignment of a participant to a particular therapeutic strategy; no additional diagnostic or monitoring procedures shall be applied to the participants; epidemiological methods shall be used for the analysis of collected data; the prescription of any medication for the treatment of the epileptic syndrome occur before the collection of the data in this study and is clearly separated from the decision to include the participant in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥2 years
* Disease history of at least 24 months from date of first seizure
* Medical history of epilepsy associated with moderate to severe intellectual disability, cognitive developmental delay or cognitive regression
* Medical history of onset of seizures in early childhood (≤ 8 years)
* Failure of adequate trials of two tolerated and appropriately chosen and used Anti-Epileptic Drug (AED) schedules (whether as monotherapies or in combination) to achieve sustained seizure freedom
* Ongoing refractory epilepsy
* MRI and EEG data are available for the participant
* Participants (or their parents/ legal representative as appropriate) have provided written informed consent / assent form to collect the data specified.

Exclusion Criteria:

* Normal cognitive development.
* Any acute symptomatic seizures in participants with underlying developmental delay.
* Any progressive intellectual and neurological deterioration conditions.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with rare epilepsy syndromes up to the date of the most recent visit at the study site.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants With and Without Diagnosis of an Epilepsy Syndrome | 5 months
  Understand the proportion of participants with and without diagnosis of an epilepsy syndrome, as described by the International League Against Epilepsy (ILAE) diagnostic manual located at https://www.epilepsydiagnosis.org/
Understand the Clinical Practice Criteria | 5 months
  Understand the clinical practice criteria used for specific syndromic diagnosis of participants with refractory epilepsy associated with developmental delay.
Clinical Practice Diagnostic Criteria Compared to ILAE | 5 months
  Compare clinical practice diagnostic criteria to those proposed by the ILAE and identify potential areas of educational need.
Understand the Time to Formal Diagnosis | 5 months
  Understand the time to diagnosis, from first seizure to formal diagnosis of a specific syndrome.
Unclassified Epilepsy | 5 months
  Evaluate if unclassified epilepsy can be grouped with common electroclinical phenotype features.

CONTACTS AND LOCATIONS:
Locations (19):
- France (3):
  - Unité de neuropédiatrie, CHU Angers, Angers
  - Department of Neurology - Foundation John Bost, La Force
  - Hospital St Louis DRCI, CHU Bicêtre, Paris
- Germany (12):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Institut der Diagnostik der Epilepsien, Berlin
  - Zentrum für Sozialpädiatrie und Neuropädiatrie (DBZ), Vivantes Klinikum, Berlin
  - Gesellschaft für Epilepsieforschung e. V., Bielefeld
  - Klinik für Epileptologie, Universitätsklinikum Bonn, Bonn
  - Klinik für Neurologie, Heilig Geist-Krankenhaus GmbH, Cologne
  - Klinik Für Kinder- und Jugendmedizin, Neuropadiatrie und Epilepsiezentrum, Frankfurt
  - Department of Neurology / Epileptology, University Medicine Greifswald, Greifswald
  - Klinik für Kinder-und Jugendmedizin II, Universitätsklinikum Schleswig-Holstein, Kiel
  - Epilepsiezentrum Kork, Kork
  - Department of Neurologie University of Magdeburg, Magdeburg
  - Abteilung für Epileptologie, ZfP Südwürttemberg, Ravensburg
- Italy (2):
  - I.R.C.C.S. Giannina Gaslini, Genova
  - Oasi Research Institute, Troina
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Ruber Internacional, Madrid